CLINICAL TRIAL: NCT04983329
Title: Systematic Quality Improvement With Realtime Event Support
Acronym: SQUIRES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Paul Kerby, Assoc Prof of Anesthesiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202107031
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Telemedicine
Keywords: Telemedicine; Quality-Improvement; surgical antibiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improvement in administration of surgical antibiotic prophylaxis. (Other): The eight-month module will include a baseline phase, educational interventions, real-time guidance from a remote telemedicine center, regular feedback regarding adherence to protocols related to that module, and continued silent monitoring.
  Interventions: Other: Telemedicine intervention

INTERVENTIONS:
Other: Telemedicine intervention — Following education, the telemedicine center will subsequently monitor operating rooms included in this trial for protocol adherence for three-months. The telemedicine center is staffed by attending anesthesiologists, resident anesthesiologists, certified registered nurse anesthetists (CRNAs) and student registered nurse anesthetists (SRNAs) and is currently providing evidence-based support to clinicians in a subset of operating rooms and post-anesthesia care unit (PACU) beds at Barnes-Jewish Hospital.

SUMMARY:
The goal of this study is to improve perioperative quality metric performance in patients receiving anesthesia care provided by Washington University Department of Anesthesiology. In this protocol, we describe (1) the use of telemedicine-augmented quality improvement interventions to enhance on-time dosage of surgical prophylactic antibiotics, while (2) carrying out large scale monitoring of surgical site infection incidence in the target population. If this quality improvement framework is found to be feasible and successful, we plan subsequently to study its application to additional perioperative quality metrics, including many pertinent to surgical site infection incidence such as perioperative glucose monitoring and management, and intraoperative temperature management.

ELIGIBILITY:
Inclusion Criteria:

* Patients having procedures at Barnes-Jewish Hospital in suites not part of the TECTONICS trial will be included.

Exclusion Criteria:

* Patients enrolled in the ongoing TECTONICS intraoperative Anesthesiology Control Tower telemedicine trial at Barnes-Jewish Hospital will be excluded from this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25506 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Improvement in administration of surgical antibiotic prophylaxis- intervention period | 3 months
  1a. Increase the rate of on-time surgical antibiotic prophylaxis administration prior to incision during the intervention period.
Improvement in administration of surgical antibiotic prophylaxis-after quality improvement intervention | 2 months
  1b. Increase the rate of on-time surgical antibiotic prophylaxis administration prior to incision six weeks after the quality improvement intervention is completed.
Improvement in administration of surgical antibiotic prophylaxis | 8 months
  1c. Increase the rate of on-time re-dosing of antibiotic prophylaxis throughout the duration of the trial.

SECONDARY OUTCOMES:
Surgical site infection rate | 8 months
  Decrease the proportion of patients which develop surgical site infections throughout the duration of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Wildes, MD, Principal Investigator — Washington Univeristy School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No